CLINICAL TRIAL: NCT06927921
Title: Assessemnt of the Knoweldge ,Attitudes and Practices of Diabetic Kidney Disease Among Diabetic Patients
Brief Title: Assessement of the Knoweldge ,Attitudes,Practices of Diabetic Kidney Disease Among Diabetic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Abdelaziz Hassan Mahmoud, Resident doctor in south valley university, Assiut University
Other Study IDs: assessment of diabetic kidney
Record Dates: First submitted 2025-03-28; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research aims to evaluate the levels of knowledge , attitudes and practices, of diabetic kidney disease among diabetic patients.

DETAILED DESCRIPTION:
Diabetic kidney disease is defined as patients with diabetes mellitus who have persistent proteinuria for at least three consecutive measurements per year, or a decrease in GFR (<90 ml/min/1.73m²) .Diabetic kidney disease is a severe microvascular complication frequently associated with both type 1 and type 2 diabetes mellitus, is a leading cause of renal failure. The condition can also lead to accelerated cardiovascular disease and macrovascular complications.

In Egypt, DM is a dilemma and a fast-expanding concern. According to the International Diabetes Federation (IDF), the prevalence of DM among Egyptian adults is 15.2%, which may be an underestimation.Public awareness, knowledge, and preventive practices are crucial in mitigating the onset and progression of diabetic nephropathy. Gaining insights into the general population's awareness, knowledge, attitudes, and practices (A-KAP) pertaining to this condition is crucial for the development of effective educational campaigns and preventative strategies.

ELIGIBILITY:
Inclusion Criteria:

* • Diabetic patients (either type 1or 2 DM ) with age above 18yrs old.

Exclusion Criteria:

* • CKD patients due to cause other than diabetes.

  * Patients who refuse participation in the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Across sectional study take anumber of diabetic patients either type 1or 2DM with age above 18yrs old to evaluate the level of knoweldge,attitudes and practices of diabetic kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
evaluation of the knowledge, attitude and practice of chronic kidney disease among the diabetic patients through a questionnaire | Baseline
  CKD screening index, which is divided into three different scales. The knowledge scale consists of 24 items regarding general knowledge of CKD, including its definition, risk factors, signs, symptoms, and complications. The attitudes scale, composed of 15 items, was used to assess the attitudes of diabetic patients toward CKD signs and symptoms and the ability to seek appropriate social and medical help related to their concerns. The practice score consists of 12 items that evaluate the health practices of each patient to prevent CKD. The validity and reliability of this screening index were examined and guaranteed and used in its arabic edition in another study .
  The correct answer was given one point, zero points for an incorrect answer, a Therefore, more correct answers meant greater knowledge of DM.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Abdelazeem Ahmed Seleem, Prof, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Assuit university, Assuit University
  - Assuit university, Asyut

REFERENCES:
- [Background] Kato M, Natarajan R. Diabetic nephropathy--emerging epigenetic mechanisms. Nat Rev Nephrol. 2014 Sep;10(9):517-30. doi: 10.1038/nrneph.2014.116. Epub 2014 Jul 8. PMID 25003613